CLINICAL TRIAL: NCT00003459
Title: Phase II Study of Antineoplastons A10 and AS2-1 In Patients With Brain Stem Glioma
Brief Title: Antineoplaston Therapy in Treating Patients With Brain Stem Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066491; BC-BT-11 (Other: Burzynski Research Institute, Inc)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Brain Stem Gliomas
Keywords: recurrent adult brain stem glioma; untreated adult brain stem glioma; untreated childhood brain stem glioma; recurrent childhood brain stem glioma
MeSH Terms: interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dosage is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with a brain stem glioma will receive Antineoplaston therapy (Atengenal + Astugenal)
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for a brain stem glioma provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of brain stem gliomas.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on children (> 6 months of age) and adults with newly-diagnosed or recurrent brain stem gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with a brain stem glioma, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with a brain stem glioma.

OVERVIEW: This is a single arm, open-label study in which patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size in measured utilizing MRI scans, which are performed every 8 weeks for the first 2 years, every 3 months for the 3rd and 4th years, every 6 months for the 5th and 6th years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed (except if medically contraindicated) brain stem glioma that is unlikely to respond to existing therapy and for which no curative therapy exists.
* Tumor must be at least 5 mm in maximum diameter

PATIENT CHARACTERISTICS:

Age:

* 6 months or greater

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other serious concomitant disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed (must be on stable dose for at least 1 week before study entry)

Radiotherapy:

* At least 8 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* No prior Antineoplaston therapy

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1996-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burzynski, S.R., Janicki, J., Burzynski, G., Marszalek, A. A Phase II Study of Antineoplastons A10 and AS2-1 in Patients with Brainstem Gliomas. The Report on Non-Diffuse Intrinsic Pontine Glioma (Protocol BT-11). Journal of Cancer Therapy, 6: 334-344, 2015
- [Background] Burzynski SR, Janicki TJ, Burzynski GS, Marszalek A. The response and survival of children with recurrent diffuse intrinsic pontine glioma based on phase II study of antineoplastons A10 and AS2-1 in patients with brainstem glioma. Childs Nerv Syst. 2014 Dec;30(12):2051-61. doi: 10.1007/s00381-014-2401-z. Epub 2014 Apr 10. PMID 24718705
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourty patients were recruited between March 1996 and January 2007. All study subjects were seen at the Burzynski Clinic in Houston, TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 40
Completed | 31 (Nine patients were not evaluable.)
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: Years] | 11.2 [3.5 to 43.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 31
Participants
  Complete Response | 5
  Partial Response | 4
  Stable Disease | 8
  Progressive Disease | 14

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 40
Percentage of participants
  6 months overall survival | 62.5
  12 months overall survival | 37.5
  24 months overall survival | 27.5
  36 months overall survival | 25.0
  48 months overall survival | 20.0
  60 months overall survival | 20.0

ADVERSE EVENTS:
Time Frame: 10 years, 9 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 25/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Hypotension (Cardiac disorders) | 1 — The hypotension was not related to Antineoplaston therapy.
Central venous catheter infection (Infections and infestations) | 4 — None of the central venous catheter infections were related to Antineoplaton therapy.
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 — The fatigue (asthenia, lethargy, malaise) was possibly related to Antineoplaston therapy.
Fever (General disorders) | 2 — Neither of the fevers were related to Antineoplaston therapy.
Dehydration (Gastrointestinal disorders) | 1 — The dehydration was not related to Antineoplaston therapy.
Diarrhea (Gastrointestinal disorders) | 1 — The diarrhea was not related to Antineoplaston therapy.
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 — The dysphagia (difficulty swallowing) was not related to Antineoplaston therapy.
Incontinence, anal (Gastrointestinal disorders) | 1 — The incontinence, anal, was not related to Antineoplaston therapy.
Leak, GI: Stomach (Gastrointestinal disorders) | 1 — The leak, GI: stomach, was not related to Antineoplaston therapy.
Nausea (Gastrointestinal disorders) | 1 — The nausea was not related to Antineoplaston therapy.
Vomiting (Gastrointestinal disorders) | 2 — Neither episode of vomiting was related to Antineoplaston therapy.
Hemorrhage, CNS (Nervous system disorders) | 4 — None of the hemorrhages, CNS, were related to Antineoplaston therapy.
Pancreatitis (Hepatobiliary disorders) | 3 — None of the pancreatitises were related to Antineoplaston therapy.
Infection (documented clinically): Blood (Infections and infestations) | 2 — None of the Infections (documented clinically): blood, were related to Antineoplaston therapy.
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 7 — None of the infections (documented clinically): lung (pneumonia), were related to Antineoplaston therapy.
Infection (documented clinically): Soft tissue NOS (Infections and infestations) | 1 — The infection (documented clinically): soft tissue NOS, was not related to Antineoplaston therapy.
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 2 — Neither of the infections (documented clinically): upper airway NOS, were related to Antineoplaston therapy.
Hypernatremia (Investigations) | 4 — Two of the four hypernatremias were possibly related to Antineoplaston therapy.
Hypocalcemia (Investigations) | 1 — The hypocalcemia was not related to Antineoplaston therapy.
Hypophosphatemia (Investigations) | 1 — The hypophosphatemia was not related to Antineoplaston therapy.
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1 — The extremity-upper (function) was not related to Antineoplaston therapy.
Confusion (Nervous system disorders) | 1 — The confusion was not related to Antineoplaston therapy.
Hydrocephalus (Nervous system disorders) | 3 — None of the hydrocephaluses were related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 4 — None of the seizures were related to Antineoplaston therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 7 — One of the somnolences/depressed levels of consciousness was possibly related to Antineoplaston therapy.
Pain: Abdomen NOS (General disorders) | 1 — The pain: abdomen NOS was not related to Antineoplaston therapy.
Pain: Head/headache (General disorders) | 1 — The pain: head/headache was not related to Antineoplaston therapy.
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 — The ARDS was not related to Antineoplaston therapy.
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 — None of the dyspneas (shortnesses of breath) were related to Antineoplaston therapy.
Thrombosis/thrombus/embolism (Vascular disorders) | 1 — The thrombosis/thrombus/embolism was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=40)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 6
Hemoglobin (Blood and lymphatic system disorders) | 15
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8
Lymphopenia (Blood and lymphatic system disorders) | 9
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7
Platelets (Blood and lymphatic system disorders) | 5
Hypertension (Cardiac disorders) | 4
Central Venous Catheter Infection (Infections and infestations) | 7
Central Venous Catheter Non-functional (General disorders) | 9
Central Venous Catheter Other (General disorders) | 4
Central Venous Catheter Pain (General disorders) | 4
Dehydration (General disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 22
Fever (General disorders) | 5
Insomnia (General disorders) | 4
Rigors/chills (General disorders) | 5
Weight gain (General disorders) | 8
Edema/Fluid retention (General disorders) | 5
Cushingoid appearance (Endocrine disorders) | 3
Diarrhea (Gastrointestinal disorders) | 13
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 4
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 16
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 21
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 4
Infection (documented clinically): Bladder (urinary) (Infections and infestations) | 4
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 4
Infection (documented clinically): Mucosa (Infections and infestations) | 7
Infection (documented clinically): Sinus (Infections and infestations) | 4
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 8
Albumin, serum-low (hypoalbuminemia) (Investigations) | 5
Hypercholesteremia (Investigations) | 6
Hyperglycemia (Investigations) | 5
Hypernatremia (Investigations) | 21
Hypocalcemia (Investigations) | 8
Hypoglycemia (Investigations) | 13
Hypokalemia (Investigations) | 33
Hypomagnesemia (Investigations) | 9
Hypophosphatemia (Investigations) | 5
Proteinuria (Investigations) | 7
SGOT (Investigations) | 9
SGPT (Investigations) | 14
Ataxia (incoordination) (Nervous system disorders) | 4
Confusion (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 5
Mood alteration: Agitation (Nervous system disorders) | 3
Neurology - Other (Nervous system disorders) | 3
Neuropathy: cranial: CN VII Motor-face; Sensory-taste (Nervous system disorders) | 3
Neuropathy: motor (Nervous system disorders) | 3
Somnolence/depressed level of consciousness (Nervous system disorders) | 20
Speech impairment (Nervous system disorders) | 5
Diplopia (Eye disorders) | 4
Pain: Abdomen NOS (General disorders) | 4
Pain: Head/headache (General disorders) | 13
Pain: Joint (General disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Incontinence, urinary (Renal and urinary disorders) | 4
Urinary frequency/urgency (Renal and urinary disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No